CLINICAL TRIAL: NCT07168317
Title: Efficacy and Safety of Tislelizumab in Combination With Cyclophosphamide, Mitoxantrone Liposomes, Chidamide, and Prednisone in the Treatment of New Diagnosed AITL: a Multicenter, Single-arm, Prospective Clinical Study
Brief Title: Tislelizumab , Cyclophosphamide, Mitoxantrone Liposomes, Chidamide, and Prednisone in the Treatment of New Diagnosed AITL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL332-01
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: New Diagnosed Angioimmunoblastic T-Cell Lymphoma
MeSH Terms: interventions — tislelizumab; Cyclophosphamide; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with new diagnosed angioblastic T cell lymphoma (Experimental): Patients with new diagnosed angioblastic T cell lymphoma
  Interventions: Drug: tislelizumab in combination with cyclophosphamide, mitoxantrone liposomes, chidamide, and prednisone

INTERVENTIONS:
Drug: tislelizumab in combination with cyclophosphamide, mitoxantrone liposomes, chidamide, and prednisone — tislelizumab: 200mg on d1 every 3 weeks; chidamide: 20mg twice a week at least 3 days apart; cyclophosphamide: 750mg/m2 on Day 1 of each cycle, every 4 weeks; mitoxantrone liposomes: 20mg/m2 on Day 1, every 4 weeks; prednisone: 100mg/day on Day 1 to Day 5 of each course, every 4 weeks.

SUMMARY:
Angioimmunoblastic T-cell lymphoma (AITL) is a rare and aggressive lymphoma. At present, the treatment of new diagnosed AITL has limited efficacy and a high recurrence rate. The study seeks to explore the possibility of improving the efficacy of immunotherapy and chemotherapy and epigenetically regulated drugs.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of AITL according to WHO classification in 2016, and pathological diagnosis of AITL according to WHO classification in 2016, and at least one evaluable or measurable lesion meeting Lugano2014 criteria: lymph node lesion, detectable lymph node length>1.5cm; non-lymph node lesion, detectable extra-nodal lesion length>1.0cm;

  * Never received systemic or local treatment including chemotherapy before;
  * Age ≥18 years old, male or female, ECOGPS≤3 points;
  * Life expectancy exceeds 3 months;
  * Follow-up conditions. Patients understand the characteristics of the disease and voluntarily join the study protocol for treatment and follow-up.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible for inclusion in this study:

  * Patients with abnormal liver and kidney function, specifically serum direct bilirubin, serum indirect bilirubin and/or alanine aminotransferase, aspartate aminotransferase and serum creatinine>2 times normal values, unless abnormal liver and kidney function is considered to be related to lymphoma;
  * Bone marrow failure, specifically defined as absolute neutrophil count (ANC)<1.5*10^9/L or platelets <75*10^9/L or Hb<90g/L, unless changes in hemogram are considered to be associated with lymphoma infiltration of the bone marrow;
  * Patients who have previously received local or systemic anti-tumor treatment;
  * Chronic heart failure with cardiac function class III or IV; or left ventricular ejection fraction <50%; or patients with the following cardiac diseases within 6 months: acute coronary syndrome; acute heart failure (Class III or IV of cardiac function class); patients with a history of clinically significant QT prolongation (>450 ms for men,>470 ms for women), ventricular tachycardia (VT), atrial fibrillation (AF), heart block, symptomatic coronary heart disease requiring medical treatment;
  * AIDS, syphilis, active B (HBV DNA>1*10^4 copies/ml) and hepatitis C;
  * Patients with other malignancies that are not effectively controlled; or with other hematological disorders (e.g. hemophilia, myelofibrosis, etc.), the investigator considers that the patient is not suitable for enrollment;
  * History of autoimmune disease, receiving immunosuppressive therapy before enrollment, immunosuppressive dose>10 mg/day or oral prednisone for more than 2 weeks;
  * Clinically uncontrolled active infection (including bacterial, fungal or viral infections), and drug therapy is ineffective;
  * Patients with uncontrolled hemophagocytic syndrome;
  * Patients who have received secondary surgery or above within 3 weeks before treatment;
  * Patients who have participated in clinical trials of other drugs within 30 days before enrollment or are participating in clinical trials of other new drugs;
  * Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
  * Known allergies to investigational drug components;
  * The investigator considers that the enrollment is not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure | Time forecasting: 24 months
  To evaluate the Objective Response Rate (Complete response+Partial response) of tirelizumab in combination with cyclophosphamide, mitoxantrone liposomes, sidaraniline, and prednisone in subjects with relapsed/refractory angioimmunoblastic T-cell lymphoma

SECONDARY OUTCOMES:
24-month Overall Survival Rate in relapsed/refractory AITL | From first dose until death from any cause (assessed at 24 months)
  Proportion of patients alive at 24 months after initiation of tirelizumab combination therapy
24-month Progression-free Survival Rate in relapsed/refractory AITL | From first dose until first documented progression or death (assessed at 24 months)
  Proportion of patients without disease progression at 24 months per Lugano 2014 criteria
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time forecasting: 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China